CLINICAL TRIAL: NCT05302141
Title: Effects of 3D Printing Assistive Device on ADL Function in Patients With Nerve Injury
Brief Title: Effects of Assistive Device on ADL Function in Patients With Nerve Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202201010
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-02

CONDITIONS: Nerve Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing assistive device group (Experimental): experimental (3D printing assistive device) groups for 4 weeks of treatment (thirty minutes a time, twice a week).
  Interventions: Behavioral: Wear 3D printing assistive device
- universal cuff groups (Active Comparator): control (universal cuff) groups for 4 weeks of treatment (thirty minutes a time, twice a week).
  Interventions: Behavioral: Wear universal cuff device

INTERVENTIONS:
Behavioral: Wear 3D printing assistive device — Wear 3D printing aids and engage in functional tasks, including eating, typing, and writing.
  At home: use daily, 30 minutes each time; Treatment room: 30 minutes twice a week
  Arms: 3D printing assistive device group
Behavioral: Wear universal cuff device — Wear universal cuff aids and engage in functional tasks, including eating, typing, and writing.
  At home: use daily, 30 minutes each time; Treatment room: 30 minutes twice a week
  Arms: universal cuff groups

SUMMARY:
Our study is aimed to evaluate the effect of 3D printing assistive device on hand function for patients with neural injury.

DETAILED DESCRIPTION:
Background: Injury to the central or peripheral nerves can lead to limited hand function and further affect the ability of daily life. The use of assistive devices can assist functional activities and reduce the phenomenon of non-use. 3D printing technology was used to construct personalized, complicated orthosis, and one piece to reduce assembly time. But the evidence most are product development, but few of study investigate the effectiveness and it cannot be widely used for hand injuries.

Aim: To evaluate the effect of 3D printing assistive device on hand function for patients with neural injury.

Methods: Thirty neural injury patients were recruited and randomized into experimental (3D printing assistive device) or control (universal cuff) groups for 4 weeks of treatment (thirty minutes a time, twice a week). The performance was assessed by a blinded assessor included Active Range of motion (AROM), Box and block test, Grip dynamometer, upper extremity task, Disability of the arm, shoulder and hand questionnaire(DASH), General Health Questionnaire(GHQ-12) and Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST). The practice performance and adverse effect were recorded. Collected data will be analyzed with nonparametric tests by SPSS version 20.0, and alpha level was set at .05.

Keywords: Neural injury, 3D printing, assistive device, hand function.

ELIGIBILITY:
Inclusion Criteria:

* The medical record shows the diagnosis of central or peripheral nerve injury, and the onset is more than three months
* Able to understand wearing operation instructions and have the ability to give informed consent
* Able to control shoulder lifting and bending elbows, but difficult to grasp tools

Exclusion Criteria:

* Older than 75 years old and younger than 20 years old
* Severe visual or hearing impairment
* Suffering from other neurological, cardiopulmonary, or musculoskeletal diseases that affect the subject to perform the actions required by this test.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Active joint range of motion of shoulder and elbow | Change from Baseline at 2 weeks and 4 weeks
  use a goniometer to measure the active joint movements of the shoulder and elbow, including shoulder flexion, abduction, external rotation , internal rotation, and elbow flexion angle.

SECONDARY OUTCOMES:
Box and block test (BBT) | Change from Baseline at 2 weeks and 4 weeks
  Assess grasping, transporting, and releasing small blocks, and count the number of blocks the individual moves 1 inch to the opposite side of the box in one minute.
Grip power | Change from Baseline at 2 weeks and 4 weeks
  use the Jamar Dynamometer (Asimow Engineering Co., CA, USA) grip strength device to test, ask the individual to bend the elbow and shoulder adduct, and hold the grip strength device firmly, and measure the average 3 times in total
Hand function tasks | Change from Baseline at 2 weeks and 4 weeks
  Complete the tasks of writing, spoon, and typing. The writing task is based on the writing sub-item of the Basic Literacy Test, and the individual is asked to write a short sentence, the content is 25 words, count the number of words in two minute; spoon task, ask the client to use a spoon to scoop five kidney beans into a can, and count the seconds it takes; one-minute typing test (https://typing.tw/), to see the number of words typed in one minute with the correct rate.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | Change from Baseline at 4 weeks
  The first and second subscales are used. To evaluate the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale., which are converted into 100 points. The higher the score, the higher the severity.
General Health Questionnaire (GHQ-12) | Change from Baseline at 4 weeks
  Self-rating scale used to measure mental health status. Respondents rated the frequency of occurrence of each item in the past month on a scale of 0 (not at all) to 3 (often). The total score can be up to 36 points, and a score of 15 or more can be defined as mental distress. The higher the score, the more serious the distress.
Daily wearing activity record sheet | Every training session during 8 sessions, total sessions continued to 4 weeks
  To record the daily wearing and practice time, the number of side effects, such as soreness, pain, injury, etc.
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | The end of the study at 4 weeks
  The questionnaire is a subjective self-administered scale for the use of assistive devices, with a 5-point scale (strongly agree to strongly disagree), including beauty, complexity, weight , resistance, comfort, easy to wear, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hsinchieh Lee, master, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amaral DS, Duarte ALBP, Barros SS, Cavalcanti SV, Ranzolin A, Leite VMM, Dantas AT, Oliveira ASCRC, Santos PS, Silva JCA, Marques CDL. Assistive devices: an effective strategy in non-pharmacological treatment for hand osteoarthritis-randomized clinical trial. Rheumatol Int. 2018 Mar;38(3):343-351. doi: 10.1007/s00296-017-3892-1. Epub 2017 Nov 28. PMID 29185087
- [Background] Armour BS, Courtney-Long EA, Fox MH, Fredine H, Cahill A. Prevalence and Causes of Paralysis-United States, 2013. Am J Public Health. 2016 Oct;106(10):1855-7. doi: 10.2105/AJPH.2016.303270. Epub 2016 Aug 23. PMID 27552260
- [Background] Baronio G, Harran S, Signoroni A. A Critical Analysis of a Hand Orthosis Reverse Engineering and 3D Printing Process. Appl Bionics Biomech. 2016;2016:8347478. doi: 10.1155/2016/8347478. Epub 2016 Aug 9. PMID 27594781
- [Background] Basteris A, Nijenhuis SM, Stienen AH, Buurke JH, Prange GB, Amirabdollahian F. Training modalities in robot-mediated upper limb rehabilitation in stroke: a framework for classification based on a systematic review. J Neuroeng Rehabil. 2014 Jul 10;11:111. doi: 10.1186/1743-0003-11-111. PMID 25012864
- [Background] Bethoux F. Spasticity Management After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):625-39. doi: 10.1016/j.pmr.2015.07.003. Epub 2015 Sep 26. PMID 26522902
- [Background] Cazon, A., Aizpurua, J., Paterson, A., Bibb, R., Campbell, R. I. J. V., & Prototyping, P. (2014). Customised design and manufacture of protective face masks combining a practitioner-friendly modelling approach and low-cost devices for digitising and additive manufacturing: This paper analyses the viability of replacing conventional practice with AM method to make customized protective face masks. 9(4), 251-261.
- [Background] Chae DS, Kim DH, Kang KY, Kim DY, Park SW, Park SJ, Kim JH. The functional effect of 3D-printing individualized orthosis for patients with peripheral nerve injuries: Three case reports. Medicine (Baltimore). 2020 Apr;99(16):e19791. doi: 10.1097/MD.0000000000019791. PMID 32311991
- [Background] Chen HM, Chen CC, Hsueh IP, Huang SL, Hsieh CL. Test-retest reproducibility and smallest real difference of 5 hand function tests in patients with stroke. Neurorehabil Neural Repair. 2009 Jun;23(5):435-40. doi: 10.1177/1545968308331146. Epub 2009 Mar 4. PMID 19261767
- [Background] Sanchez-Lopez Mdel P, Dresch V. The 12-Item General Health Questionnaire (GHQ-12): reliability, external validity and factor structure in the Spanish population. Psicothema. 2008 Nov;20(4):839-43. PMID 18940092
- [Background] Diment LE, Thompson MS, Bergmann JH. Three-dimensional printed upper-limb prostheses lack randomised controlled trials: A systematic review. Prosthet Orthot Int. 2018 Feb;42(1):7-13. doi: 10.1177/0309364617704803. Epub 2017 Jun 24. PMID 28649911
- [Background] Fitzpatrick, A. P., Mohanned, M. I., Collins, P. K., & Gibson, I. (2017). Design of a patient specific, 3D printed arm cast. KnE Engineering, 135-142.
- [Background] Funch A, Kruse NB, la Cour K, Peoples H, Waehrens EE, Brandt A. The association between having assistive devices and activities of daily living ability and health-related quality of life: An exploratory cross-sectional study among people with advanced cancer. Eur J Cancer Care (Engl). 2019 May;28(3):e13002. doi: 10.1111/ecc.13002. Epub 2019 Feb 10. PMID 30740805
- [Background] Gerhardt JJ, Rondinelli RD. Goniometric techniques for range-of-motion assessment. Phys Med Rehabil Clin N Am. 2001 Aug;12(3):507-27. PMID 11478185
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Harman, D., & Craigie, S. J. E. G. M. (2011). Gerotechnology series: Toileting aids. 2(5), 314-318.
- [Background] Hepherd, R. J. E. G. M. (2011). Aids for bathing and showering. 2(3), 190-193.
- [Background] Hunzeker, M., & Ozelie, R. (2021). A Cost-Effective Analysis of 3D Printing Applications in Occupational Therapy Practice. The Open Journal of Occupational Therapy, 9(1), 1-12.
- [Background] Janson R, Burkhart K, Firchau C, Hicks K, Pittman M, Yopps M, Hatfield S, Garabrant A. Three-dimensional printed assistive devices for addressing occupational performance issues of the hand: A case report. J Hand Ther. 2020 Apr-Jun;33(2):164-169. doi: 10.1016/j.jht.2020.03.025. Epub 2020 May 16. PMID 32423845
- [Background] Jumani, M., Shaikh, S., & Shah, S. A. J. S. I. (2014). RAPID MANUFACTURING TECHNIQUE FOR FABRICATION OF CUSTOM-MADE FOOT ORTHOSES. 26(1).
- [Background] Keller M, Guebeli A, Thieringer F, Honigmann P. Overview of In-Hospital 3D Printing and Practical Applications in Hand Surgery. Biomed Res Int. 2021 Mar 26;2021:4650245. doi: 10.1155/2021/4650245. eCollection 2021. PMID 33855068
- [Background] Lee KH, Kim DK, Cha YH, Kwon JY, Kim DH, Kim SJ. Personalized assistive device manufactured by 3D modelling and printing techniques. Disabil Rehabil Assist Technol. 2019 Jul;14(5):526-531. doi: 10.1080/17483107.2018.1494217. Epub 2018 Oct 14. PMID 30318956
- [Background] Liang HW, Wang HK, Yao G, Horng YS, Hou SM. Psychometric evaluation of the Taiwan version of the Disability of the Arm, Shoulder, and Hand (DASH) questionnaire. J Formos Med Assoc. 2004 Oct;103(10):773-9. PMID 15490028
- [Background] Long TM, Woolverton M, Perry DF, Thomas MJ. Training needs of pediatric occupational therapists in assistive technology. Am J Occup Ther. 2007 May-Jun;61(3):345-54. doi: 10.5014/ajot.61.3.345. PMID 17569392
- [Background] Lubbes, E. (2016). Investigation and Assessment of Upper-Limb Prosthetic Care and Business Model Design for 3D-Printed Prostheses in the Netherlands.
- [Background] Ma HI, Hwang WJ, Tsai PL, Hsu YW. The effect of eating utensil weight on functional arm movement in people with Parkinson's disease: a controlled clinical trial. Clin Rehabil. 2009 Dec;23(12):1086-92. doi: 10.1177/0269215509342334. PMID 19906764
- [Background] Marque P, Gasq D, Castel-Lacanal E, De Boissezon X, Loubinoux I. Post-stroke hemiplegia rehabilitation: evolution of the concepts. Ann Phys Rehabil Med. 2014 Nov;57(8):520-529. doi: 10.1016/j.rehab.2014.08.004. Epub 2014 Aug 23. PMID 25282582
- [Background] Martin, L. M. J. A. J. o. O. T. (1988). Clinical Mechanics of the Hand. 42(3), 199-199.
- [Background] McDonald SS, Levine D, Richards J, Aguilar L. Effectiveness of adaptive silverware on range of motion of the hand. PeerJ. 2016 Feb 15;4:e1667. doi: 10.7717/peerj.1667. eCollection 2016. PMID 26893960
- [Background] Nam HS, Seo CH, Joo SY, Kim DH, Park DS. The Application of Three-Dimensional Printed Finger Splints for Post Hand Burn Patients: A Case Series Investigation. Ann Rehabil Med. 2018 Aug;42(4):634-638. doi: 10.5535/arm.2018.42.4.634. Epub 2018 Aug 31. PMID 30180536
- [Background] Nordin N, Xie SQ, Wunsche B. Assessment of movement quality in robot- assisted upper limb rehabilitation after stroke: a review. J Neuroeng Rehabil. 2014 Sep 12;11:137. doi: 10.1186/1743-0003-11-137. PMID 25217124
- [Background] Phillips, B., Zingalis, G., Ritter, S., & Mehta, K. (2015). A review of current upper-limb prostheses for resource constrained settings. Paper presented at the 2015 IEEE global humanitarian technology conference (GHTC).
- [Background] Portnova AA, Mukherjee G, Peters KM, Yamane A, Steele KM. Design of a 3D-printed, open-source wrist-driven orthosis for individuals with spinal cord injury. PLoS One. 2018 Feb 22;13(2):e0193106. doi: 10.1371/journal.pone.0193106. eCollection 2018. PMID 29470557
- [Background] Radomski, M. V., & Latham, C. A. T. (2014). Occupational therapy for physical dysfunction(7 th ed): Lippincott Williams & Wilkins.
- [Background] Roda-Sales A, Vergara M, Sancho-Bru JL, Gracia-Ibanez V, Jarque-Bou NJ. Effect on hand kinematics when using assistive devices during activities of daily living. PeerJ. 2019 Oct 8;7:e7806. doi: 10.7717/peerj.7806. eCollection 2019. PMID 31608177
- [Background] Sari MI, Sahin I, Gokce H, Oksuz C. Ring orthosis design and production by rapid prototyping approach. J Hand Ther. 2020 Apr-Jun;33(2):170-173. doi: 10.1016/j.jht.2019.02.003. Epub 2019 Apr 10. PMID 30981658
- [Background] Saunders, R., Astifidis, R., Burke, S. L., CHT, M., Higgins, J., & McClinton, M. A. (2015). Hand and upper extremity rehabilitation: a practical guide: Elsevier Health Sciences.
- [Background] Skymne C, Dahlin-Ivanoff S, Claesson L, Eklund K. Getting used to assistive devices: ambivalent experiences by frail elderly persons. Scand J Occup Ther. 2012 Mar;19(2):194-203. doi: 10.3109/11038128.2011.569757. Epub 2011 May 2. PMID 21534712
- [Background] Somers, M. F. (2001). Spinal cord injury: functional rehabilitation: Prentice Hall.
- [Background] Stowe, S., Hopes, J., & Mulley, G. J. E. g. m. (2010). Gerotechnology series: 2. Walking aids. 1(2), 122-127.
- [Background] Takla, M. K., Mahmoud, E. A., & Abd El-Latif, N. J. B. o. F. o. P. T. (2018). Jebsen Taylor Hand Function test: Gender, dominance, and age differences in healthy Egyptian population. 23(2), 85-93.
- [Background] Thibaut A, Chatelle C, Ziegler E, Bruno MA, Laureys S, Gosseries O. Spasticity after stroke: physiology, assessment and treatment. Brain Inj. 2013;27(10):1093-105. doi: 10.3109/02699052.2013.804202. Epub 2013 Jul 25. PMID 23885710
- [Background] Toth, L., Schiffer, A., Nyitrai, M., Pentek, A., Told, R., & Maroti, P. (2020). Developing an anti-spastic orthosis for daily home-use of stroke patients using smart memory alloys and 3D printing technologies. Materials & Design, 195, 109029.
- [Background] Yoo HJ, Lee S, Kim J, Park C, Lee B. Development of 3D-printed myoelectric hand orthosis for patients with spinal cord injury. J Neuroeng Rehabil. 2019 Dec 30;16(1):162. doi: 10.1186/s12984-019-0633-6. PMID 31888695